CLINICAL TRIAL: NCT04397965
Title: Cascade CGM 15-Day US Performance Assessment
Brief Title: Cascade Continuous Glucose Monitor (CGM) 15-Day US Performance Assessment
Acronym: CUSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: WaveForm Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: EXT-1040
Record Dates: First submitted 2020-04-02; First posted 2020-05-21 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-05

CONDITIONS: Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental: Continuous Monitoring (Experimental): Intervention: Device: Cascade Continuous Glucose Monitoring System
  Interventions: Device: Cascade Continuous Glucose Monitor

INTERVENTIONS:
Device: Cascade Continuous Glucose Monitor — Continuous Glucose Monitoring
  Other Names: Cascade CGM

SUMMARY:
To assess a 15-day wear period of the Cascade Continuous Glucose Monitoring (CGM) System

DETAILED DESCRIPTION:
To assess a 15-day wear period for the Cascade CGM. The study wear period includes four in-clinic days in which frequent blood draws and Yellow Springs Instrument (YSI) glucose measurements will be performed. Participants will be blinded to CGM glucose values during the study. A retrospective performance assessment will be conducted following the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 or type 2 (on insulin therapy) diabetes mellitus for at least 6 months
* 18 years of age or older
* Currently self-monitoring capillary blood glucose (on average at least three times per day or more) or using a CGM for at least three months -Willing to follow all study procedures, including attending all clinic visits (including in- clinic sessions during which a venous line will be inserted for blood sampling), wearing a CGM sensor(s) for fifteen days, performing fingertip glucose tests for self-monitoring, and keeping a diary of activities.
* Be willing to wear 2 investigational CGM devices.

Exclusion Criteria:

1. Known allergy to medical grade adhesives
2. Magnetic Resonance Imaging (MRI) scheduled during fifteen-day CGM sensor wear period
3. Persons with type 2 diabetes using diet and exercise only for diabetes management
4. Used an investigational drug within 30 days prior to study entry
5. Hematocrit < 35% for females and <40% for males (obtained during screening)
6. Inadequate veins (in the opinion of the investigator) or known contraindication to placement of a dedicated peripheral line for venous blood withdrawal
7. Symptomatic coronary artery disease with a history of angina, or history of a myocardial infarction or coronary intervention (e.g., percutaneous transluminal coronary angioplasty (PTCA), stent placement), or coronary artery bypass graft (CABG) within the past six months
8. Diagnosis of the following diabetic autonomic neuropathies: orthostatic hypotension, heart rate anomalies, gastroparesis
9. Cerebrovascular incident within the past six months
10. History or presence of eczema, psoriasis, atopic or contact dermatitis
11. Subject must not be pregnant at the start of the study.
12. Current use or within one-week exposure to topical medications at the proposed insertion sites
13. Seizure disorder (epilepsy)
14. Malignancy within the past five years, except basal cell or squamous cell skin cancers
15. Major surgical operation within 30 days prior to screening
16. Other medical conditions that would pose safety concerns, interfere with study conduct or seriously compromise study integrity (reason for exclusion will be clearly documented by investigator or designee)
17. Subject has experienced severe hypoglycemia or severe hyperglycemia in the last six months. Severe hypoglycemia is defined as having low blood glucose levels that requires assistance from another person to treat. Severe hypoglycemia is classed as a diabetic emergency. Severe hyperglycemia is defined as a blood ketone level >1.6 millimolar (mM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Use | 15 days
  Validate the feasibility of a 15-day wear period of the Cascade CGM. The primary endpoint is an 80% sensor survival rate over a 15-day wear period, which includes four in-clinic days and eleven at-home days.

SECONDARY OUTCOMES:
Performance | 15 days
  Accuracy performance compared to YSI readings. The secondary endpoints are: to achieve <15% Mean Average Relative Difference (MARD) and <20mg/dL Mean Average Difference (MAD) compared to YSI readings during the four in-clinic days and to assess Blood Glucose Meter (BGM) fingerstick calibration success.

IPD SHARING:
Plan to Share IPD: No